CLINICAL TRIAL: NCT02032602
Title: Efficacy of Dry Needling on Myofascial Trigger Points in Adults Over 65 Years Old With Non-specific Shoulder Pain: Single Blind Randomized Controlled Clinical Trial
Brief Title: Dry Needling on Myofascial Trigger Points in Older Adults With Nonspecific Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cesar Calvo Lobo, PT, MSc, doctoral student, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v5EGIU
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Shoulder Pain
Keywords: Myofascial Pain Syndromes; Trigger Point; Shoulder Pain; Aged
MeSH Terms: conditions — Shoulder Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, CG: Active MTrP (Active Comparator): a single session of physical therapy intervention which will be consisted on Deep Dry Needling of the active MTrP most hyperalgesic to palpation of the infraspinatus muscle homolateral to painful shoulder
  Interventions: Other: Deep Dry Needling
- 2, EG: Active+Latent MTrPs (Experimental): The same treatment described above for the Control Group, combined with the Deep Dry Needling of the most hyperalgesic latent MTrP, both located in the infraspinatus muscle homolateral to the painful shoulder.
  Interventions: Other: Deep Dry Needling

INTERVENTIONS:
Other: Deep Dry Needling

SUMMARY:
Background: Non-specific shoulder pain has a high prevalence in older adults and provokes functional alterations. Besides, there are difficulties for its clinical diagnosis, lack of effectiveness in the treatment and not much evidence is found regarding invasive physical therapy techniques in this population.

Purpose: To determine the efficacy of a single physical therapy intervention with deep dry needling on latent and active myofascial trigger points in older adults with non-specific shoulder pain.

Methods: Pilot Study, Single Blind Randomized Controlled Clinical Trial on 60 subjects aged 65 and over, will be diagnosed with nonspecific shoulder pain. The study will be approved by the Clinical Research Ethics Committee of the area. Sample will be recruited at their home and at a care center, and randomly will be distributed in Experimental Group (n=30), which will be received a session of Deep Dry Needling on an active and a latent Myofascial Trigger Points of the infraspinatus muscle; and Control Group (n=30), receiving a session of Deep Dry Needling only on an active Myofascial Trigger Point. A blind examiner will be evaluated Pain Intensity, Pain Pressure Threshold (anterior deltoid; extensor carpi radialis brevis) and Grip Strength, before, immediately after intervention and after a week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* people aged 65 or over with uni or bilateral non-specific shoulder pain and with at least one active and one latent MTrP in the infraspinatus homolateral to the painful shoulder

Exclusion Criteria:

* prior diagnosis of myopathy or neuropathy; cognitive deficit in the medical record; cervical spine, rotator cuff tendons or glenohumeral joint problems in the medical record; corticoid infiltration or local anaesthetic during the previous year or during follow-up; surgical procedure affecting the upper limb or preceding cervical; ingestion of antiaggregant, anti-coagulant, analgesic or anti-inflammatory medication or abusive substances in the week prior to treatment and during follow-up were excluded from the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain Intensity on the Numerical Rating Scale (NRS) at 5 minutes | Baseline, 5 minutes
  Pain Intensity was measured with the Numerical Rating Scale (NRS) of 11 points (interval of 0-10), where 0 corresponds to no pain and 10 corresponds to the worst pain imaginable. In order to show a parametric analysis of the obtained data, a graphical representation of 11 spaces describes levels for the discrimination of the patient. The subjects will be asked to determine the subjective pain intensity of the painful shoulder using a finger.
Change from baseline in Pain Pressure Threshold of anterior deltoid at 5 minutes | Baseline, 5 minutes
  Pressure Pain Threshold (PPT) will be measured with a WAGNER FDK/FDN Series Force Dial Fisher type analogue algometer (Wagner Instruments, Greenwich, USA) which varies between 0-10 kg/cm2. After indicating the most hyperalgesic latent Myofascial Trigger Point (MTrP) of anterior deltoid muscle (located in referred pain area and with the same C5-6 segmentary innervation levels), examiner will determine PPT of such point.
Change from baseline in Maximum Grip Strength at 5 minutes | Baseline, 5 minutes
  Maximum grip strength, defined as the maximum isometric muscular force in kg used in the manual pressure of a hydraulic dynamometer, will be measured with a JAMAR type hydraulic manual analogical dynamometer with an interval of 0-90kg to objectify the weakness of latent Myofascial Trigger Points (MTrPs) of the forearm. According to the fatigability of older adults, a single measurement will be performed to measure the manual grip strength.
Change from baseline in Pressure Pain Threshold of extensor carpi radialis brevis at 5 minutes | Baseline, 5 minutes
  Pressure Pain Threshold (PPT) will be measured with a WAGNER FDK/FDN Series Force Dial Fisher type analogue algometer (Wagner Instruments, Greenwich, USA) which varies between 0-10 kg/cm2. After indicating the most hyperalgesic latent Myofascial Trigger Point (MTrP) of extensor carpi radialis brevis muscle (located in referred pain area and with the same C5-6 segmentary innervation levels), examiner will determine PPT of such point.
Change from baseline in Pain Intensity on the Numerical Rating Scale (NRS) at 1 week | Baseline, 1 week
  Pain Intensity was measured with the Numerical Rating Scale (NRS) of 11 points (interval of 0-10), where 0 corresponds to no pain and 10 corresponds to the worst pain imaginable. In order to show a parametric analysis of the obtained data, a graphical representation of 11 spaces describes levels for the discrimination of the patient. The subjects will be asked to determine the subjective pain intensity of the painful shoulder using a finger.
Change from baseline in Pressure Pain Threshold of anterior deltoid at 1 week | Baseline,1 week
  Pressure Pain Threshold (PPT) will be measured with a WAGNER FDK/FDN Series Force Dial Fisher type analogue algometer (Wagner Instruments, Greenwich, USA) which varies between 0-10 kg/cm2. After indicating the most hyperalgesic latent Myofascial Trigger Point (MTrP) of anterior deltoid muscle (located in referred pain area and with the same C5-6 segmentary innervation levels), examiner will determine PPT of such point.
Change from baseline in Maximum Grip Strength at 1 week | Baseline, 1 week
  Maximum grip strength, defined as the maximum isometric muscular force in kg used in the manual pressure of a hydraulic dynamometer, will be measured with a JAMAR type hydraulic manual analogical dynamometer with an interval of 0-90kg to objectify the weakness of latent Myofascial Trigger Points (MTrPs) of the forearm. According to the fatigability of older adults, a single measurement will be performed to measure the manual grip strength.
Change from baseline in Pressure Pain Threshold of extensor carpi radialis brevis at 1 week | Baseline, 1 week
  Pressure Pain Threshold (PPT) will be measured with a WAGNER FDK/FDN Series Force Dial Fisher type analogue algometer (Wagner Instruments, Greenwich, USA) which varies between 0-10 kg/cm2. After indicating the most hyperalgesic latent Myofascial Trigger Point (MTrP) of extensor carpi radialis brevis muscle (located in referred pain area and with the same C5-6 segmentary innervation levels), examiner will determine PPT of such point.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcala, Alcalá de Henares, Madrid, Spain